CLINICAL TRIAL: NCT04825600
Title: Diagnosis of Toxoplasma Gondii Infection by Exploration of Cellular Immunity
Brief Title: Diagnosis of Toxoplasma Gondii Infection by Exploration of Cellular Immunity (TOXCELL)
Acronym: TOXCELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-AOI-07
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Toxoplasmosis; Toxoplasma Infections; Toxoplasmosis, Congenital; Toxoplasmosis Recurrent
MeSH Terms: conditions — Toxoplasmosis; Toxoplasmosis, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- toxo+ (Other)
  Interventions: Diagnostic Test: anti-Toxoplasma gondii IgG and IgM dosage; Diagnostic Test: cellular test
- uninfected (Other)
  Interventions: Diagnostic Test: anti-Toxoplasma gondii IgG and IgM dosage; Diagnostic Test: cellular test
- mother and child duo (Other)
  Interventions: Diagnostic Test: anti-Toxoplasma gondii IgG and IgM dosage; Diagnostic Test: cellular test
- toxo+ more than 10 years (Other)
  Interventions: Diagnostic Test: anti-Toxoplasma gondii IgG and IgM dosage; Diagnostic Test: cellular test

INTERVENTIONS:
Diagnostic Test: anti-Toxoplasma gondii IgG and IgM dosage — blood sample performed to check the toxoplasma serological diagnosis
Diagnostic Test: cellular test — blood sample performed to evaluate the anti T. gondii cellular immunity and to compare results to the toxoplasma serological diagnosis

SUMMARY:
Toxoplasmosis is a parasitic disease caused by Toxoplasma gondii and transmitted to humans through the consumption of raw or undercooked infected meat and / or by poorly washed vegetables. It can be transmitted from the pregnant woman to the fetus when infection occurs during pregnancy leading to congenital toxoplasmosis. Once infected, it is considered that the subject harbors cyst forms of the parasite in the muscles and brain for life with a risk of reactivation when immunocompromised. Recently, questions have been raised about the persistence of these cysts.

Currently, only serological diagnosis can demonstrate the infection. This is done by detecting IgM and IgG directed against the parasite. Although humoral immunity is useful to diagnose toxoplasmosis, the cellular immunity is responsible of the main protective role during infection with the secretion of cytokines such as gamma interferon. In some situations, the serological diagnosis is limited: in immunocompromised subjects, some immunocompetent patients, in children with congenital toxoplasmosis, in which the anti T. gondii antibodies are no longer detectable. In order to have a true evaluation of the capacities of the immune system of each individual against T. gondii infection, it is necessary to evaluate the effector immune cells.

The main objective of this protocol is to set up a cellular test with the stimulation of lymphocyte by T. gondii. For this objective, 20 subjects (10 positive, 10 negative for Toxoplasmosis serology) will be included. The secondary objective will be to compare the cellular diagnosis (evaluation by ELISA of the secretion of gamma interferon in the supernatant of cells stimulated by the Ag) with the serological diagnosis (IgG and IgM Alinity Abbott and Western blot LD Bio) in 3 groups of 10 patients: chronically infected patients, uninfected patients, patients with congenital toxoplasmosis as well as to assess the persistence or not of cellular and humoral immunity against T. gondii in 10 patients who had acute toxoplasmosis with a known date infection more than 10 years. Thus, 60 patients will be included for a total study period of 24 months.

This study will thus allow the sponsor to have a clear understanding whether a subject is able or not to react against T. gondii infection.

DETAILED DESCRIPTION:
Toxoplasmosis is a parasitic disease caused by Toxoplasma gondii and transmitted to humans through the consumption of raw or undercooked infected meat and / or by poorly washed vegetables. It can be transmitted from the pregnant woman to the fetus when infection occurs during pregnancy leading to congenital toxoplasmosis. Once infected, it is considered that the subject harbors cyst forms of the parasite in the muscles and brain for life with a risk of reactivation when immunocompromised. Recently, questions have been raised about the persistence of these cysts.

Currently, only serological diagnosis can demonstrate the infection. This is done by detecting IgM and IgG directed against the parasite. Although humoral immunity is useful to diagnose toxoplasmosis, the cellular immunity is responsible of the main protective role during infection with the secretion of cytokines such as gamma interferon. In some situations, the serological diagnosis is limited: in immunocompromised subjects, some immunocompetent patients, in children with congenital toxoplasmosis, in which the anti T. gondii antibodies are no longer detectable. In order to have a true evaluation of the capacities of the immune system of each individual against T. gondii infection, it is necessary to evaluate the effector immune cells.

The main objective of this protocol is to set up a cellular test with the stimulation of lymphocyte by T. gondii. For this objective, 20 subjects (10 positive, 10 negative for Toxoplasmosis serology) will be included. The secondary objective will be to compare the cellular diagnosis (evaluation by ELISA of the secretion of gamma interferon in the supernatant of cells stimulated by the Ag) with the serological diagnosis (IgG and IgM Alinity Abbott and Western blot LD Bio) in 3 groups of 10 patients: chronically infected patients, uninfected patients, patients with congenital toxoplasmosis as well as to assess the persistence or not of cellular and humoral immunity against T. gondii in 10 patients who had acute toxoplasmosis with a known date infection more than 10 years. Thus, 60 patients will be included for a total study period of 24 months.

The patients included must be over 15 years of age, unknown HIV (questionnaire), not immunocompromised (questionnaire), with a known T. gondii serological status, affiliated with social security and having signed the informed consent form. Patients with known immunosuppression or immunosuppressive therapy (questionnaire) will be included.

The patients thus selected will be included in the study. This study will allow the sponsor to acquire knowledge of the real immunity of the patients, if they harbor cysts with a risk of reactivation in case of immunosuppression and, for pregnant women known with congenital toxoplasmosis, whether lymphocytes from these women are able to react against T. gondii.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 15 years of age, for minor patients signature of both parents or parent authority representative
* Unknown HIV (questionnaire)
* Non-immunocompromised (questionnaire)
* Known serological status with toxoplasmosis
* Social Security Affiliate
* Informed Consent Signature

Exclusion Criteria:

* Presence of known immunosuppression or immunosuppressive therapy (questionnaire).
* HIV-positive people will be excluded due to the immunosuppressive action of HIV

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
Implement a cell test with lymphocytic stimulation by toxoplasmic antigen and screening for T. gondii infection to assess cellular immunity against T. gondii | 12 months
  to develop the cell test locally and optimize it. Cell immunity will be evaluated by assay of gamma interferon secretion in the supernatant of patient cells stimulated by parasitic antigen. For this, we will carry out the Toxoféron set up in Lyon and we will compare its realization to from the globular cap and from a ficoll that allows to select the cells of immunity.

SECONDARY OUTCOMES:
Compare cell diagnosis with serological diagnosis and assess whether or not cellular and humoral immunity against T. gondii. | 24 months
  will perform cellular tests and serological diagnosis. Serological diagnosis will be made by the detection of IgG and IgM anti Toxoplasmic by chemiluminescence (ABBOTT reagent on automaton ALINITY i) and by the realization of Western Blot confirmation TOXO LDBIO II. The subject will be considered positive for serological antibody diagnosis if he has positive or doubtful IgG and a Western blot positive..

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No
no data sharing plan is schedule